CLINICAL TRIAL: NCT00309595
Title: A Multi-Center Prospective, Randomized, Two-Arm Clinical Investigation of the Cordis SMARTTM Nitinol Self Expandable Stent Versus Balloon Angioplasty Only for the Treatment of Superficial Femoral Artery Occlusions.
Brief Title: The Study to Compare SMART Nitinol Stent and Balloon Angioplasty
Acronym: SIT-UP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Dr. Hans-Peter Stoll - Medical Affairs Director, Cordis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EE04-03
Record Dates: First submitted 2006-03-31; First posted 2006-04-03 (Estimated); Last update posted 2009-06-12 (Estimated); Status verified 2009-06

CONDITIONS: Superficial Femoral Artery Occlusions
MeSH Terms: interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Cordis SMART™ nitinol self expandable stent
  Interventions: Device: stent
- 2 (Active Comparator): balloon
  Interventions: Device: balloon

INTERVENTIONS:
Device: stent — Cordis SMART™ Nitinol Stent System
  Arms: 1
Device: balloon — balloon angioplasty
  Arms: 2

SUMMARY:
This is a multi-center prospective, randomized, two-arm study evaluating performance of the Cordis SMART™ Nitinol Stent System compared to balloon angioplasty. Patients will be randomized on a 1:1 basis. It is anticipated that a total of 120 patients will be entered into the study.

Objective of the study is: Performance of the Cordis S.M.A.R.T.™ (CONTROL™) Nitinol Stent System for the treatment of superficial femoral artery (SFA) long de novo or restenotic lesions (≥ 70% stenosis or occlusions) in comparison with balloon angioplasty as determined by Binary Restenosis (≥50% restenosis based on a peak systolic velocity ratio ≥ 2.5) at one year as demonstrated by Duplex sonography.

DETAILED DESCRIPTION:
The study population will consist of 120 symptomatic peripheral vascular disease patients with SFA occlusions. The disease will consist of symptomatic, de novo or restenotic occlusions (5 - 22 cm) on diagnostic imaging. The occlusions must not extend beyond the proximal popliteal artery. For the purpose of this protocol, no lesion within 3 cm of the upper part of the patella may be treated. At least one calf vessel must be patent. Reference vessel diameter must be >= 4.0 to <= 6.0 mm.

Trial participants who meet all entry criteria, will be randomized to the SMART™ Nitinol Stent or balloon angioplasty.

Patients will be followed for 12 months after the procedure. Study examinations will be done at screening, procedure time, discharge, 1, 6 and 12 months after the study procedure.

This study will be conducted as an investigator initiated multicenter study with 6 study centers in Switzerland. Principal investigators will be Prof. Amann, PD Dr. med T. Pfammatter (University Hospital Zürich) and Prof. I. Baumgartner, Prof. J. Triller (University Hospital Bern).

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic leg ischemia by Rutherford Classification (category 1, 2, 3, 4 or 5); duration of intermittent claudication (category 1-3) should be at least 3 months;
2. One de-novo or restenotic SFA with an occluded length > 5 to < 22 cm;
3. Patent popliteal artery on the index side (without > 50% stenotic (re) stenotic lesions) and at least single vessel infrapopliteal runoff (without > 50% stenotic (re) stenotic lesions). However, balloon angioplasty to further improve the blood flow is allowed at the index procedure.

Exclusion Criteria:

1. Revascularization involving the same limb 30 days prior to the index procedure or a planned revascularization within 30 days after the index procedure;
2. Patients having severe stenoses or total occlusions of the iliac artery on the same side must be excluded. However, intervention to restore adequate blood flow during the index procedure (prior to the treatment of the target lesion) is allowed;
3. Requiring stent placement in the popliteal artery. For the purpose of this protocol all lesions are to be located at least three centimetres proximal to the superior edge of the patella.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Binary restenosis by Duplex Ultrasound. | 1 year

SECONDARY OUTCOMES:
Technical success defined as a successful access and deployment of the device with recanalization. | at the time of deployment
Procedural complications. | up to the moment the catheter sheath introducer has been removed
Procedural success as defined by successful recanalization, without the occurence of a Serious Adverse Event (SAE). | up to the catheter sheath introducer has been removed
Occurrence of Adverse events (AE) and Serious Adverse Events (SAE) in-hospital. | 1, 6 and 12 months
Ankle Brachial Index (ABI). | discharge, 1, 6 and 12 months
Restenosis measured by Duplex sonography. | 1, 6 and 12 months
Target Lesion revascularisation (TLR). | 1 year
Target Vessel revascularisation (TVR). | 1 year
Target Limb revascularisation. | 1 year
The number of revascularisations in both limbs. | 1 year
Clinical categorization of chronic limb ischemia by means of the Rutherford classification. | 1, 6 and 12 months
Pain free and absolute walking distance (treadmill testing) as compared to baseline testing. | 1 and 12 months post index procedure
Amputation of the index limb. | 1 year
Cardiovascular events (ACS, TIA, stroke, vascular death). | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Iris Baumgartner, MD, Principal Investigator — Leitende Aerztin & Leiterin Vaskuläre Forschung - University Hospital Bern; Beatrice Amann, MD, Principal Investigator — Leitende Ärztin Angiologie - University Hospital Zurich
Locations (2):
- Switzerland (2):
  - Univeristy Hospital Bern, Bern
  - University Hospital Zurich, Zurich